CLINICAL TRIAL: NCT06127810
Title: A Pilot Study of Gadopiclenol for Imaging Central Nervous System (CNS) Tumors at Point of Care Magnetic Resonance Imaging (MRI)
Brief Title: MRI Gadopiclenol Enhanced Imaging of CNS Tumors
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor backed out of the trial.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00129735
Record Dates: First submitted 2023-10-30; First posted 2023-11-13 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Image
Keywords: MRI; Radiology
MeSH Terms: interventions — gadopiclenol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- 3T Contrast Enhanced Images First
  Interventions: Device: CE MRI on 0.064T Scanner; Drug: Gadopiclenol
- 0.064 Contrast Enhanced Images First
  Interventions: Device: CE MRI on 0.064T Scanner; Drug: Gadopiclenol

INTERVENTIONS:
Device: CE MRI on 0.064T Scanner — Pt will undergo contrast enhanced images using Gadopiclenol on Hyperfine MRI
Drug: Gadopiclenol — Subjects will receive Gadopiclenol instead of standard of care contrast

SUMMARY:
The purpose of this pilot study is to compare a standard of care MRI scan to a non-standard of care MR imaging with portable (0.064 Tesla) MRI following the administration of non-SOC contrast called Gadopiclenol on 10 subjects with known brain tumors.

Participants will be randomized to receive either standard MRI or portable MRI first following contrast injection

DETAILED DESCRIPTION:
This study compares a routine MRI scan with a new portable MRI scanner known as the "Hyperfine" using a contrast dye called Gadopiclenol, the contrast is FDA approved. If participants choose to participate in this study, they will receive two MRI scans on the same day. One on the traditional standard of care MRI scanner and the other on the new portable Hyperfine MRI. The Hyperfine MRI scanner is not FDA approved due to being a very low risk medical device. However, the device is compliant with all of the FDA requirements regarding design control regulations and risk analysis. Participants will only receive one contrast injection that will be used for both scans. The selection of which scan is given first will be randomly selected (50/50 chance). Participation in this study will last two days. The first day participants will receive both MRI scans and the second day participants will receive a phone call from the research staff to check on them.

ELIGIBILITY:
Inclusion Criteria

* Female or male adult patient (18 years and older).
* Patient presenting, at the time of inclusion, with known or highly suspected focal areas of disrupted Blood Brain Barrier (BBB) due to primary or secondary tumor/s. This lesion must have been detected on a previous imaging procedure (computerized Tomography (CT) or MRI).
* Patient scheduled for a routine CNS contrast-enhanced MRI examination for clinical reasons.
* Patient able and willing to participate in the study.
* Patient with health insurance.

Exclusion Criteria

* Patient presenting with acute or chronic Grade III (at least) renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m² based on eGFR assessment on the day of each MRI.
* Pregnant or breast-feeding female patient (a female patient of childbearing potential must be using a medically approved contraception method until the last study visit).
* Patient with any contraindication to MRI examinations including active implants, passive implants which are MRI incompatible, and metallic foreign bodies.
* Patient with known contra-indication(s) to the use or with known sensitivity to any GBCA.
* Patient having received any contrast agent (MRI or CT) within 3 days prior to study gadopiclenol administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting, at the time of inclusion, with known or highly suspected focal areas of disrupted Blood Brain Barrier (BBB) due to primary or secondary tumor/s.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Visibility of lesions | 1 Day
  Visibility of lesions and diagnostic capabilities of 0.068T MRI